CLINICAL TRIAL: NCT07204340
Title: An Open-Label, Multicenter, Phase 1 Trial to Evaluate the Safety, Pharmacokinetics, and Anti-Tumor Activity of TLN-372 as a Single Agent and in Combination With Other Anti-Tumor Agents, in Patients With Advanced KRAS Mutant Solid Tumors
Brief Title: TLN-372 in Advanced KRAS Mutant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Treeline Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TLN-372-2501
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: KRAS Mutant Solid Tumors
Keywords: KRAS mutant solid tumors; KRAS
MeSH Terms: interventions — Cetuximab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Agent (Experimental)
  Interventions: Drug: TLN-372
- Combination Treatment (Experimental)
  Interventions: Drug: TLN-372 in combination with cetuximab; Drug: TLN-372 in combination with pembrolizumab

INTERVENTIONS:
Drug: TLN-372 — Specified dose on specified days
  Arms: Single Agent
Drug: TLN-372 in combination with cetuximab — Specified dose on specified days
  Arms: Combination Treatment
Drug: TLN-372 in combination with pembrolizumab — Specified dose on specified days
  Arms: Combination Treatment

SUMMARY:
The primary purpose of this study is to evaluate the safety, pharmacokinetics, and anti-tumor activity of TLN-372 as a single agent and in combination with other anti-tumor agents, in patients with advanced KRAS mutant solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have measurable disease at study entry.
2. Patients must have locally advanced or metastatic KRAS mutant solid tumors.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Adequate organ function.

Exclusion Criteria:

1. Patients must not have active brain metastases.
2. Patients must not have current or past history of central nervous system (CNS) involvement.
3. Patients must not have major surgery or severe trauma within 4 weeks prior to the start of the study.
4. Patients must not have any condition, including significant acute or chronic medical illness, active or uncontrolled infection, or the presence of laboratory abnormalities, that places patients at unacceptable risk of participating in this study.
5. Patients must not have clinically significant cardiovascular disease.
6. Pregnant or lactating.
7. Conditions that could affect drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2031-12-03 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing adverse events (AEs) that meet protocol-defined dose-limiting toxicity (DLT) criteria following administration of TLN-372 | Up to 2 years
Incidence and severity of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse Events (TRAEs) leading to dose modification and discontinuation. | Up to 2 years
Anti-tumor activity of TLN-372 by evaluating the objective response rate (ORR) according to the RESIST v1.1 | Up to 2 years

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of TLN-372 | Up to 2 years
Time to peak drug concentration (Tmax) of TLN-372 | Up to 2 years
Minimum observed plasma concentration (Cmin) of TLN-372 | Up to 2 years
Area Under the Plasma Concentration-Time Curve (AUC) of TLN-372 | Up to 2 years
Anti-tumor activity of TLN-372 by evaluating the duration of response (DOR) as assessed by the time from the date of first objective response to the date of disease progression | Up to 2 years
Frequency of dose interruptions, reductions and dose intensity | Up to 2 years
Clinically significant ECG QT Interval from baseline in safety laboratory test results, assessed as per NCI CTCAE v5.0 | Up to 2 years
Clinically significant laboratory abnormalities from baseline in safety laboratory test results, assessed as per NCI CTCAE v5.0 | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Washington University Medical Campus, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No